CLINICAL TRIAL: NCT04066166
Title: Accuracy of Rib Palpation for Dry Needling of Deep Periscapular Musculature, Measured With Ultrasound
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Daniel Cushman, Principle Investigator, University of Utah
Other Study IDs: 0084226
Record Dates: First submitted 2019-08-12; First posted 2019-08-26 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Trigger Point Pain, Myofascial
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Palpation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects: Healthy
  Interventions: Diagnostic Test: Palpation

INTERVENTIONS:
Diagnostic Test: Palpation — All healthy subjects palpated

SUMMARY:
Ultrasound was used to identify the location of a rib. This was compared to a practitioner's ability to palpate the area.

DETAILED DESCRIPTION:
Ultrasound was used to identify the location of a rib. This was compared to a practitioner's ability to palpate the area. The purpose of this study is to identify if practitioners are as accurate as they think they are in identifying ribs. This is important, as mis-identifying a rib may put patients at risk for inadvertent needle entry into the lung.

ELIGIBILITY:
Inclusion Criteria:

* Anyone with ribs

Exclusion Criteria:

* No children

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All healthy participants
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Accuracy | 1 year
  Number of participants who were appropriately identified compared to ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cushman, Principal Investigator — UNIVERSITY OF UTAH ORTHOPAEDICS CENTER

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-06-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT04066166/Prot_SAP_000.pdf
  • Informed Consent Form (2015-06-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT04066166/ICF_001.pdf